CLINICAL TRIAL: NCT03773835
Title: A Single-center, Open-label, Uncontrolled, and Dose-escalation Study Evaluating Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Single IV Dose of HSK3486 Injectable Emulsion in Healthy Subjects.
Brief Title: A Study Evaluating Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Single IV Dose of HSK3486 Injectable Emulsion in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-101
Record Dates: First submitted 2018-12-06; First posted 2018-12-12 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2016-08

CONDITIONS: Anesthesia; Sedation
MeSH Terms: interventions — HSK3486

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSK3486 (Experimental): 0.15mg/kg, 0.40mg/kg, 0.60mg/kg, 0.90mg/kg,
  Interventions: Drug: HSK3486

INTERVENTIONS:
Drug: HSK3486 — Mmanual IV bolus injection completed in 1 minute.

SUMMARY:
his single-center, open-label, uncontrolled, and dose-escalation study evaluated the safety, tolerability, and pharmacokinetics/pharmacodynamics of single IV dose of HSK3486 injectable emulsion in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females with full capacity for civil conduct, between 18 and 49 years old (inclusive);
2. Body weight > 45 kg, and body mass index (BMI) ≥ 19 and ≤24 kg/m2;
3. Blood pressure between 90-140/60-90 mmHg; heart rate between 60-99 bpm; body temperature between 35.8-37.5 ºC; respiration rate between 12-24 breaths per minute; SpO2 when inhaling > 95%;
4. Normal physical examination, laboratory tests (blood routine, blood biochemistry, and urine routine), 12-Led ECG, posteroanterior and lateral chest x-ray, and or abnormal but without clinical significance (determined by investigator); no potential difficult airway;
5. Subjects must understand the procedures and methods of this study, and be willing to provide informed consent and to complete the trial in strict accordance with clinical trial protocol.

Exclusion Criteria:

1. Known sensitivity to propofol, excipient in propofol medium and long chain fat emulsion injection, excipient in HSK3486 injectable emulsion;
2. contraindicated in general anesthesia;
3. Received any one of the following medications or treatments prior to screening/enrollment:

   1. History of medication abuse or any signs of chronic benzodiazepines use (such as insomnia, anxiety, spasms) within 3 months prior to screening, or a positive urine medication test (during screening or at baseline);
   2. Participated in clinical trials involving any medications or medical devices within 3 months prior to screening, or participated in 3 or more drug clinical trials within the past year;
4. History or evidence of increased risk of sedation or anesthesia, such as cardiovascular disease, respiratory disease, cerebrovascular disease, gastrodintestinal disease and other system disease prior to the screening and/or baseline period;
5. Laboratory results that meet any of the following during screening/enrollment:

   1. Positive for HBsAg, HCV, or HIV;
   2. Abnormal hepatic or renal function confirmed after re-examination;

      * ALT or AST > ULN;
      * Creatinine > ULN;
6. History of smoking for more than 3 weeks and/or respiratory irritation caused by smoking within 3 months prior to screening;
7. History of alcohol abuse within 3 months prior to screening or a positive alcohol test (baseline);
8. Women who are pregnant or breastfeeding; women of child-bearing potential or men who are unwilling to use contraception during the trial;
9. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Apnea | First dose of study drug on day 1
  No movement of chest wall and cessation of end-tidal carbon dioxide waveform > 15 seconds.
Safety by measurement of Adverse Events | First dose of study drug on day 1

SECONDARY OUTCOMES:
Modified observer's assessment of alertness/sedation（MOAA/S） | From first dose of study drug until fully alert on day 1
  Observe the change of modified observer's assessment of alert /sedation during the whole trial
Bispectral index （BIS） | From first dose of study drug until fully alert on day 1
Median effective dose (ED50) | From first dose of study drug until fully alert on day 1
Peak concentration (Cmax) | From the start of administration to 48 hours after administration
Time to plasma peak concentration(Tmax) | From the start of administration to 48 hours after administration
Terminal elimination half life (t1/2z) and mean residence time (MRT) | From the start of administration to 48 hours after administration
Mean residence time (MRT) | From the start of administration to 48 hours after administration
Area Under the Curve (AUC0-30min, AUC0-1h, AUC0-last, and AUC0-inf) | From the start of administration to 48 hours after administration
Total clearance (CL) | From the start of administration to 48 hours after administration